CLINICAL TRIAL: NCT07276074
Title: Evaluation of the Relevance of Antithrombin Prescriptions at Strasbourg University Hospitals
Acronym: EPPATHUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9308
Record Dates: First submitted 2025-03-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Antithrombinemia
Keywords: Anticoagulants; Antithrombinemia; Extracorporeal membrane oxygenation; Renal replacement therapy; Cardiopulmonary bypass

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antithrombin (AT) is a physiological inhibitor of the coagulation cascade. In therapeutics, its presence in sufficient quantities is necessary for the pharmacological activity of unfractionated heparin (UFH) and partially low-molecular-weight heparin (LMWH).

In intensive care, patients are mostly treated with anticoagulants for either preventive or curative purposes, particularly for those whose care requires renal replacement therapy (RRT), extracorporeal membrane oxygenation (ECMO), or cardiopulmonary bypass (CPB). The use of various types of membranes associated with these procedures can lead to degradation of blood proteins (including AT). An imbalance in hemostasis can then occur, resulting in ineffective anticoagulation. At the Strasbourg University Hospitals (HUS), these medications are directly available in the intensive care units, allowing for immediate administration in an emergency. Pharmaceutical and medical analysis is therefore not performed before administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥18 years old)
* Female and male
* Having received antithrombin during the study period, in intensive care or operating room during the period from January 1, 2022 to December 31, 2023.

Exclusion Criteria:

* Subject (and/or their legal representative, if applicable) having expressed their opposition to the reuse of their data for scientific research purposes
* Minor subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult subject (≥18 years old) having received antithrombin during the study period, in intensive care or operating room during the period from January 1, 2022 to December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overview of antithrombin prescriptions | Up to 1 year
  This is a retrospective study describing antithrombin prescriptions at the Strasbourg University Hospitals over a one-year period (from January 1, 2022 to December 31, 2023)

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie et Réanimation chirurgicale - CHU de Strasbourg - France, Strasbourg, France